CLINICAL TRIAL: NCT00054990
Title: The Effects Of Antiepileptic Drugs On Cortical Excitability
Brief Title: Effects of Antiepileptic Drugs on Brain Excitability
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 030107; 03-N-0107
Record Dates: First submitted 2003-02-15; First posted 2003-02-17 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-03

CONDITIONS: Healthy
Keywords: Antiepileptic Drugs; Cortical Excitability; Transcranial Magnetic Stimulation; Epilepsy; TMS; Healthy Volunteer; HV
MeSH Terms: conditions — Epilepsy

SUMMARY:
This study will evaluate the usefulness of transcranial magnetic stimulation (TMS) in measuring cortical excitability. The cortex is the outer part of the brain. Patients with seizures have increased cortical excitability and are often treated with antiepileptic drugs to reduce this excitability. The therapeutic effects of antiepileptic drugs are usually tracked with blood tests that measure their blood levels. However, these blood tests may not always correctly reflect the effects of the drugs on the brain.

TMS has been used successfully to measure cortical excitability in many neurological diseases, including epilepsy, and may be helpful in measuring drug effects on the brain directly. For this procedure, a wire coil is held over the scalp. A brief electrical current is passed through the coil, creating a magnetic pulse that stimulates the brain. This may cause a pulling sensation on the skin under the coil and twitching in muscles of the face, arm, or leg. During the stimulation, the participant may be asked to tense certain muscles slightly or perform other simple actions.

Healthy normal volunteers between 18 and 55 years of age may be eligible for this study. Candidates will be screened with a medical history, physical and neurological examination, electroencephalogram (EEG), and blood tests.

On the first day of the study, participants will have a baseline TMS and will be randomly assigned to take one of two antiepileptic drugs: group A will take the carbamazepine; group B will take lamotrigine. If they wish, participants may be admitted to the NIH Clinical Center for the first 5 days of drug administration while the proper dosage is being determined. They will then be discharged and continue taking the drug for a total of 36 days. During this time, they will have daily blood tests and TMS from days 2 through 5, and again on days 12 and 36. Group A will have additional blood sampling and TMS on days 37, 39, 44, and 53; Group B will have blood tests and TMS on days 38, 40, 45, and 53.

DETAILED DESCRIPTION:
Objectives. Epilepsy is a condition characterized by abnormally increased cortical excitability, and antiepileptic drugs (AEDs) control epilepsy by reducing cortical excitability. Serum blood levels presently represent the standard measure utilized to track the therapeutic effects of AEDs. However, peripheral blood levels do not always reflect brain levels, or provide direct information on cortical excitability. Transcranial magnetic stimulation (TMS) is a non-invasive technique that allows accurate measures of this parameter. The purpose of this protocol is to test the hypothesis that TMS measures of cortical excitability will correlate with serum blood levels of AEDs, and reflect clinical effects on cortical function directly in healthy volunteers. This information is crucial to reach the ultimate goal of developing a reliable quantitative measurement of central physiological effects of AEDs in epileptic patients.

Study Population. 40 normal volunteers aged 18 to 55 years will be recruited for this study.

Design. Subjects will be assigned to either of two groups, with each group receiving one of the following drugs; carbamazepine (CBZ), and lamotrigine (LTG). Measures of cortical excitability will be performed using TMS in various drug treatment phases: at baseline (before drug intake); during the AED induction period (once a day for the first 5 days), after 12 days of drug intake at the maximum dose during steady state; and 3, 7, and 14 half-lives after, and finally three weeks after abrupt drug withdrawal. Blood sampling for drug levels will be performed at each TMS study.

Outcome Measures. The primary outcome variables will be MEP size, measured from recruitment curves. MEP size difference from baseline will be compared to the serum drug level for each drug.

ELIGIBILITY:
INCLUSION CRITERIA:

Normal volunteers will be male or female, aged 18 to 55 at protocol entry without any of the exclusion criteria described below.

EXCLUSION CRITERIA:

Patients will be excluded from this study if they:

1. are pregnant (tested with urine pregnancy test).
2. have severe coronary disease.
3. have metal anywhere in the cranium except the mouth.
4. have intracardiac lines.
5. have increased intracranial pressure as expressed by the presence of papilledema.
6. have cardiac pacemakers.
7. take neuroleptic or antidepressant medications.
8. any neurologic disease including epilepsy.
9. taking any psychiatric drugs.
10. any other documented systemic illness.
11. history of drug allergy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2003-02; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Burstein AH, Horton RL, Dunn T, Alfaro RM, Piscitelli SC, Theodore W. Lack of effect of St John's Wort on carbamazepine pharmacokinetics in healthy volunteers. Clin Pharmacol Ther. 2000 Dec;68(6):605-12. doi: 10.1067/mcp.2000.111530. PMID 11180020
- [Background] Cantello R, Civardi C, Cavalli A, Varrasi C, Tarletti R, Monaco F, Migliaretti G. Cortical excitability in cryptogenic localization-related epilepsy: interictal transcranial magnetic stimulation studies. Epilepsia. 2000 Jun;41(6):694-704. doi: 10.1111/j.1528-1157.2000.tb00230.x. PMID 10840401
- [Background] Chen R, Samii A, Canos M, Wassermann EM, Hallett M. Effects of phenytoin on cortical excitability in humans. Neurology. 1997 Sep;49(3):881-3. doi: 10.1212/wnl.49.3.881. PMID 9305361